CLINICAL TRIAL: NCT00988559
Title: A Pilot Study of pnGVL4a-CRT/E7 (Detox) for the Treatment of Patients With HPV16+ Cervical Intraepithelial Neoplasia 2/3 (CIN2/3)
Brief Title: Therapeutic Vaccination for Patients With HPV16+ Cervical Intraepithelial Neoplasia (CIN2/3)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: J0866; P50CA098252 (NIH); 1R21CA128232 (NIH); NA_00020850 (Other: JHM IRB)
Record Dates: First submitted 2009-10-01; First posted 2009-10-02 (Estimated); Results first posted 2018-07-09 (Actual); Last update posted 2018-07-09 (Actual); Status verified 2018-07

CONDITIONS: HPV16 Positive; Cervical Intraepithelial Neoplasia (CIN 2/3)
Keywords: high grade cervical dysplasia; treatment vaccine; therapeutic; HPV; DNA vaccine; gene therapy; gene gun; pre-cancerous
MeSH Terms: conditions — Uterine Cervical Dysplasia | interventions — Vaccines; Vaccines, DNA; Conization; Imiquimod

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- PMED Delivery - groups 1 and 2 (Experimental): Subjects will receive pNGVL4a-CRT/E7(detox) via gene gun at weeks 0, 4, 8 prior to therapeutic resection of their lesion at week 15.
  Interventions: Biological: DNA vaccination; Device: Gene gun vaccine; Procedure: therapeutic resection of the lesion
- IM injections - groups 5 and 6 (Experimental): Subjects will receive pNGVL4a-CRT/E7(detox) intramuscularly at weeks 0, 4, 8 prior to therapeutic resection of their lesion at week 15.
  Interventions: Biological: DNA vaccination; Biological: intramuscular vaccination; Procedure: therapeutic resection of the lesion
- Intralesional delivery - group 3 and 4 (Experimental): Subjects will receive pNGVL4a-CRT/E7(detox) intra-mucosally at weeks 0, 4, 8 prior to therapeutic resection of their lesion at week 15.
  Interventions: Biological: DNA vaccination; Biological: intra-lesional vaccine administration; Procedure: therapeutic resection of the lesion
- Intralesional delivery + imiquimod - group 7 (Experimental): Subjects will receive pNGVL4a-CRT/E7(detox) intra-mucosally and imiquimod applied to the cervix at weeks 0, 4, 8 prior to therapeutic resection of their lesion at week 15.
  Interventions: Biological: DNA vaccination; Biological: intra-lesional vaccine administration; Procedure: therapeutic resection of the lesion; Drug: imiquimod

INTERVENTIONS:
Biological: DNA vaccination — vaccination with pNGVL4a-CRT/E7(detox)
  Other Names: Therapeutic vaccine
Device: Gene gun vaccine — 8 micrograms (group 1) or 16 micrograms (group 2)
  Other Names: PMED administration; ND10 device
  Arms: PMED Delivery - groups 1 and 2
Biological: intramuscular vaccination — 1mg (group 3) or 3mg (group 4) of pNGVLra-CRT/E7(detox) administered intramuscularly
  Other Names: DNA vaccine
  Arms: IM injections - groups 5 and 6
Biological: intra-lesional vaccine administration — 1mg (group 5) or 3mg (group 6) of pNGVL4a-CRT/E7(detox)administered intra-lesionally
  Other Names: Intra-lesional DNA vaccination
  Arms: Intralesional delivery + imiquimod - group 7; Intralesional delivery - group 3 and 4
Procedure: therapeutic resection of the lesion — at week 15, all residual lesions will be resected
  Other Names: LEEP or cold knife conization
Drug: imiquimod — imiquimod applied to the cervix by the physician
  Arms: Intralesional delivery + imiquimod - group 7

SUMMARY:
This study will test the efficacy and safety of different routes of administration of a DNA vaccine in patients with HPV16+ CIN2/3. Subjects will be enrolled in one of six treatment groups. Subjects enrolled in the first two groups will receive vaccination intradermally with a needle-free delivery device. Subjects enrolled in groups 3 and 4 will receive vaccination intramuscularly. Subjects enrolled in groups 5 and 6 will receive vaccine intralesionally.

DETAILED DESCRIPTION:
Primary Objectives

* To evaluate the feasibility and toxicity of vaccination in women with CIN2/3 caused by HPV16
* To evaluate the effect of vaccination on histology
* To compare immunogenicity of three different routes of administration: intradermal (ID), intramuscular (IM), intralesional (IL).

Secondary Objectives:

* To evaluate changes in HPV viral load
* To evaluate the cellular immune response to vaccination
* To evaluate the humoral immune response to vaccination
* To evaluate local tissue immune response
* To correlate measures of immune response with clinical response
* To correlate measures of immune response with those observed in the preclinical model

ELIGIBILITY:
Inclusion Criteria:

* patients with high grade cervical intraepithelial lesions (CIN2/3)
* patients whose lesions are HPV16+
* patients who are age 18 or older
* patients who are able to give informed consent
* patients who are immunocompetent
* patients who are not pregnant, committed to using adequate contraception if of childbearing age
* patients who have a minimum hemoglobin level of 9

Exclusion Criteria:

* Patients with cytologic evidence of glandular dysplasia
* Patients with cytologic evidence of adenocarcinoma in situ
* Patients who are pregnant
* Patients with an active autoimmune disease
* Patients who are taking immunosuppressive medication
* Patients with concurrent malignancy except for nonmelanoma skin lesions
* Patients who have an allergy to gold.
* Patients with any evidence of damaged skin, or moles, scars, tattoos or marks at the proposed site(s) of administration that might interfere with the interpretation of local skin reactions.
* History or evidence of a physician-diagnosed chronic or recurrent inflammatory skin disease (e.g. psoriasis, eczema, atopic dermatitis, hypersensitivity) at the proposed site of administration in the past 5 years.
* Patients who have an active autoimmune disease or history of autoimmune disease requiring medical treatment with systemic immunosuppressants, including: inflammatory bowel disease, systemic vasculitis, scleroderma, psoriasis, multiple sclerosis, hemolytic anemic, or immune thrombocytopenia, rheumatoid arthritis, SLE, and Sjogren's syndrome, sarcoidosis. Asthma or COPD that does not require systemic corticosteroids or routine use of inhaled steroids is acceptable
* Patients who have received prior chrysotherapy (administration of gold salts to treat rheumatoid arthritis).
* Patients with a history of arterial or venous thrombosis
* Patients with non-healed wounds.
* Patients with a history of keloid formation ( ID delivery group only)
* Patients with a history of hepatitis B with persistent infection.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2009-09; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cornelia L Trimble, MD, Principal Investigator — Johns Hopkins University
Locations (3):
- United States (3):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Johns Hopkins Outpatient Center, Baltimore, Maryland
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 132 subjects signed consents to be screened for eligibility
  * 93 subjects signed consents, but did not meet the eligibility criteria to start the study (screen failures)
  * 39 subjects were assigned to a treatment group in the study
Period: Overall Study
Arm/Group | PMED Delivery - Groups 1 and 2 | IM Injections - Groups 5 and 6 | Intralesional Delivery - Group 3 and 4 | Intralesional Delivery + Imiquimod - Group 7
Started | 10 | 11 | 11 | 7
Completed | 9 | 9 | 9 | 6
Not Completed | 1 | 2 | 2 | 1
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 1
Not completed — Pregnancy | 0 | 1 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Participants enrolled in the study who received at least one study intervention
Groups:
- Total: Total of all reporting groups
Arm/Group | PMED Delivery - Groups 1 and 2 | IM Injections - Groups 5 and 6 | Intralesional Delivery - Group 3 and 4 | Intralesional Delivery + Imiquimod - Group 7 | Total
Number analyzed (Participants) | 10 | 11 | 11 | 7 | 39
Age, Continuous [Median (Full Range); unit: years] | 25.5 [20 to 44] | 26 [21 to 35] | 26 [23 to 35] | 26.14 [24 to 29] | 25.91 [20 to 44]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 11 | 7 | 39
  Male | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 5 | 2 | 4 | 11
  White | 9 | 5 | 9 | 3 | 26
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Related Serious Adverse Events
Description: Presence of intervention-related serious adverse events as defined by CTCAE
Time Frame: 9 months
Population: Related Serious Adverse Events
Measure: Count of Participants; unit: Participants
Arm/Group | PMED Delivery - Groups 1 and 2 | IM Injections - Groups 5 and 6 | Intralesional Delivery - Group 3 and 4 | Intralesional Delivery + Imiquimod - Group 7
Number analyzed (Participants) | 10 | 11 | 11 | 7
Participants | 0 | 0 | 0 | 0

2. Secondary Outcome: Absence of CIN2/3 Lesion by Week 15
Description: Number of participants with no CIN2/3 lesion at the week 15 visit
Time Frame: 15 weeks
Population: Number of participants who had no CIN2/3 at the week 15 resection
Measure: Count of Participants; unit: Participants
Arm/Group | PMED Delivery - Groups 1 and 2 | IM Injections - Groups 5 and 6 | Intralesional Delivery - Group 3 and 4 | Intralesional Delivery + Imiquimod - Group 7
Number analyzed (Participants) | 9 | 9 | 9 | 6
Participants | 2 | 3 | 3 | 1

ADVERSE EVENTS:
Time Frame: 41 weeks
Arm/Group | PMED Delivery - Groups 1 and 2 | IM Injections - Groups 5 and 6 | Intralesional Delivery - Group 3 and 4 | Intralesional Delivery + Imiquimod - Group 7
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/11 | 0/11 | 0/7
Other Adverse Events (participants affected / at risk) | 10/10 | 11/11 | 10/11 | 7/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PMED Delivery - Groups 1 and 2 (N=10) | IM Injections - Groups 5 and 6 (N=11) | Intralesional Delivery - Group 3 and 4 (N=11) | Intralesional Delivery + Imiquimod - Group 7 (N=7)
Injection site reactions (General disorders) | 8 (43) | 6 (10) | 1 (1) | 0 (0) — Local injection site reactions
General pain, fever, malaise/fatigue (General disorders) | 8 (44) | 8 (38) | 8 (41) | 7 (37) — Abdominal discomfort, cramping, fatigue, flu like symptoms, headaches, muscle/joint aches, nausea, pain, pruritus
Depression (Psychiatric disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Limb numbness (Nervous system disorders) | 1 (5) | 1 (1) | 0 (0) | 0 (0)
Rash (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Vaginal bleeding/spotting (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (6) — vaginal bleeding or spotting
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No